CLINICAL TRIAL: NCT03275012
Title: Randomized, Double-blind, Placebo Controlled, Superiority Phase II Study to Evaluate the Safety, Pharmacokinetic, Efficacy of Gabapentin as add-on to Morphine in Children From 3 Months to Less Than 18 Years
Brief Title: Efficacy and Safety Study of Gabapentin as add-on to Morphine in Paediatric Patients Affected by Chronic Pain
Acronym: GABA-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not started
Sponsor: Pharmaceutical Research Management srl (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-004897-40
Record Dates: First submitted 2017-08-30; First posted 2017-09-07 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Gabapentin; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Gabapentin + Morphine
  Interventions: Drug: Gabapentin + Morphine
- Group 2 (Placebo Comparator): Placebo + Morphine
  Interventions: Drug: Placebo + Morphine

INTERVENTIONS:
Drug: Gabapentin + Morphine — Gabapentin: liquid oral formulation (syrup) - 75 mg/ml-three times daily. The starting dose during the optimization period will be defined according to 2 weight groups (5-15kg and >15kg). Dose will be scaled at Day 1,3,5,14,and 21 according to a specific schedule. Maintenance dosing will be scheduled in accordance to the body weight.
  Morphine: background therapy as oral, liquid and solid formulations. Patients with BW≤30kg :liquid oral formulation four times daily throughout the whole treatment period. Patients with BM>30kg : immediate release solid and/or liquid oral formulation four times daily during titration phase and an extended release solid oral formulation twice daily during the maintenance period.
  Arms: Group 1
Drug: Placebo + Morphine — Placebo liquid oral formulation. Morphine: background therapy as oral, liquid and solid formulations. Patients with BW≤30kg :liquid oral formulation four times daily throughout the whole treatment period. Patients with BM>30kg : immediate release solid and/or liquid oral formulation four times daily during titration phase and an extended release solid oral formulation twice daily during the maintenance period.
  Arms: Group 2

SUMMARY:
The objective of the study is to evaluate the efficacy of gabapentin as adjunctive therapy to morphine in the treatment of severe chronic neuropathic or mixed pain in children from 3 months to less than 18 years of age assessed by the difference in average pain scores between treatment arms at the end of the treatment period.

DETAILED DESCRIPTION:
This paediatric trial has the objective to make gabapentin available for children with severe chronic neuropathic or mixed pain. This study will be conducted in full conformance with the ethical principles outlined in the Declaration of Helsinki, consistent with ICH-GCP (including ICH Topic E11 guideline) and applicable regulatory requirements including the Paediatric Recommendations (CE/2008).

Gabapentin has been successfully used to treat neuropathic pain in adults. In absence of specific paediatric studies it is not approved for the same condition in children.

The paediatric use of gabapentin is hampered by: a) the lack of a suitable paediatric formulation, b) the significant variability of gabapentin PK profile and c) efficacy and safety data in this specific population.

GABA-2 is a superiority trial designed to assess the potential benefit of gabapentin oral solution in augmenting the analgesic effect of morphine in children affected by severe chronic pain thus preventing or decreasing opioid tolerance, as it has been reported to happen in adults. Thus GABA-2 study is an randomized, double blind, placebo controlled, multi-centre study to evaluate the efficacy of gabapentin added to morphine in paediatric patients suffering from severe chronic pain (neuropathic or mixed with ascertained neuropathic component). The trial will include 66 patients aged from 3 months to less than 18 years affected by severe chronic neuropathic or mixed pain and in need of morphine.

Children from 3 months to <3 years of age will participate to GABA-2 on the basis of the nature of the underlying disease suggestive of a neuropathic component.

A block randomisation will be applied to assign children to gabapentin and morphine (intervention group) or gabapentin placebo and morphine (control group) in a 1:1 ratio.

Randomisation will be stratified by age-group as follows:

* 3 months - < 3 years;
* 3 years - < 8 years;
* 8 years - < 18 years.

Recruitment will start with patients ≥ 3 years of age. Patients < than 3 years of age will be recruited when results from the ongoing non-clinical toxicological study in juvenile rats will confirm the safety of gabapentin in the age subset 3 months-3 years.

The protocol has been designed to ensure double-blind conditions at randomisation and throughout the treatment period. Blinding (children, caregiver, outcome assessor) will be ensured by elaborating an identical (matching) gabapentin placebo.

The study comprises 3 stages over 18 to 22 weeks: 1st stage ( screening period of 1 week, wash out phase of max 3 days and baseline assessment of 3 days ), 2nd stage ( treatment period including an optimization phase of 3 weeks and 12 weeks of maintenance), 3rd stage (study taper lasting from 0 to 4 weeks and 1 week follow up).

The proposed formulation of the IMP test is a liquid oral formulation (syrup) containing 75 mg/ml of gabapentin. The IMP comparator is the placebo. The background therapy is morphine presented as immediate and extended-release tablets and a liquid, oral formulation. Every participant will be administered morphine and the active product or placebo.

For both study drugs, dosing will initiate at a starting dose in mg/kg/day and will be increased according to a predefined matrix to a maximum dose in mg/kg/day. Dosing will be flexibly optimised in order to maximise the potential benefits while minimising risk of AEs. There will be a maximum of 5 possible dose adjustments during the 3 weeks optimisation period.

Dosing for gabapentin during the optimization period will be defined according to two weight groups (5-15kg and >15kg). Current dosing schedule for gabapentin is the following:

* Day 1 starting dose in mg/kg/day;
* Day 3 2 times the starting dose in mg/kg/day;
* Day 5 3 times the starting dose in mg/kg/day;
* Day 14 2 times the dose of Day 5 in mg/kg/day;
* Day 21 3 times the dose of Day 5 in mg/kg/day.

Dosing of morphine is largely based on the "WHO guidelines on the pharmacological treatment of persisting pain in children with medical illnesses", 2012. The guidelines recommended starting dose for immediate release formulation of morphine are '80-200 mcg/kg every 4 hours for infants and 200-500 mcg/kg in 6 divided doses in older children. ' However, due to compliance issues a four times daily regimen (q.i.d) will be used during the titration phase of this protocol for children with body weight >30kg and throughout this study for patients with <30kg body weight.

The morphine starting dose in this study reflects the lower end of the WHO recommendation with a titration scheduled to reach a maximum daily dose of 1.2 mg/kg/day. Patients < 30kg BW will have the liquid morphine formulation, 4 times daily throughout the study and patients > 30kg will receive immediate release tablet 4 times daily, during the titration phase and extended release tablets 2 times daily during the maintenance phase.

All subjects that are completing the study or are withdrawn early must be tapered off of the gabapentin. At the visit of Early Termination or End Of Study visit, subjects will be dispensed a taper dose based on their current dose level (the dose of the medicinal product taken during the maintenance period) and should follow the dose tapering as described in the protocol.

Concomitant use of some medications that could interfere with the study will be prohibited. Unrestricted use of paracetamol and/or ibuprofen alone or in combination will be used as rescue therapy any time the patient experiences pain (pain level >4/10 measured with age- appropriate pain scales FLACC, FPS-R or NRS-11) This study includes pharmacokinetic analysis to establish a population pharmacokinetic model adequate to describe the time-course and variability of plasma concentrations of gabapentin and gabapentin plus morphine following repeat dosing in children with chronic pain.

The study includes also an optional exploratory pharmacogenomics study which requires a separate Informed Consent if the parent of the subject agrees to participate. The aims of the exploratory pharmacogenomic research is to better understand inherited genetic factors and their association with clinical assessments, which may include pharmacokinetics of gabapentin, relative susceptibility to drug-drug interactions, predisposition to side effects, and/or patients' response to treatment with gabapentin.

The study foresees also an exploratory metabolomic study that may provide insight in the mechanism of neuropathic pain and the inter-individual variation in drug response.

During this study, it is expected that a maximum of 15.9 mL of blood will be taken from every subject (male and female). Additional 2.0 ml of blood will be required from females of child bearing age for pregnancy testing.

The primary analysis of efficacy will be conducted using ANCOVA with baseline average pain score as a covariate.

The study will be conducted under the supervision of an independent Data Safety Monitoring Committee (DSMC).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 3 months to less than 18 years at screening (V1)
2. Informed consent by parent(s) and/or legal guardian according to each country legal requirement.
3. Assent, where applicable, according to each country legal requirement.Informed (co-) consent of child, where applicable, according to each country legal requirement.
4. Subjects that meet the diagnostic criteria for neuropathic or mixed pain.
5. Subjects that present with chronic pain defined as the recurrent or continuous pain persisting more than 3 months.
6. Subject that present with severe pain as defined by average pain intensity of ≥7 /10 as assessed during a 3-day screening period
7. Stable underlying disease condition and treatment.
8. Patients with Chemotherapy Induced Peripheral Neuropathy, when in clinical remission or maintenance phase of their therapeutic protocol.

Exclusion Criteria:

1. Pain duration of more than 5 years.
2. Current use of gabapentin.
3. Current use of strong opioids (morphine, methadone, fentanyl, ketamine, oxycodone).
4. History of failure to respond to adequate treatment by gabapentin or opioids for neuropathic pain.
5. History of epileptic condition (except febrile seizure disorder).
6. Subjects with diagnosis of sickle cell disease.
7. Subjects that present significant cognitive impairment.
8. Subjects that present current, controlled or uncontrolled, co-morbid psychiatric diagnosis that can impair pain diagnosis and assessment such as severe depressive conditions or psychosis.
9. Subjects with history of or current suicidal ideation or behaviour.
10. Subjects with history of substance abuse in particular opioids.
11. Subjects under prohibited concomitant medication .
12. Subjects with a body mass index (BMI) for age and gender of < 5th percentile or > 95th percentile (charts provided as Appendix 3).
13. Subjects with significant renal impairment, i.e., glomerular filtration rate < 90 mL/min/1.73 m2 (Revised Schwarz equation).
14. Subjects with significant hepatic impairment or with Aspartate Transaminase (AST) or Alanine Transaminase (ALT) enzymes 3 times the upper limit of the age-specific reference range.
15. Subjects in need for corticosteroid oral treatment or corticosteroid infiltrations to treat pain caused by infiltration or compression of neural structures, e.g. peripheral nerves or spinal cord.
16. Subjects with clinically relevant abnormal ECG at the screening visit in the discretion of the Investigator/cardiologist.
17. Subjects with known allergy, hypersensibility or clinically significant intolerance to gabapentin or any component found in the study drugs.
18. Subjects with fructose intolerance, diabetes, glucose-galactose malabsorption or lactase-isomaltase deficiency.
19. Subjects participating in another clinical interventional trial.
20. Subjects scheduled for surgery or in recovery from surgery occurring within 3 months of baseline assessment.
21. Female subjects who are pregnant or currently lactating.
22. Subjects that failed screening or were previously enrolled in this study
23. Patients with Chemotherapy Induced Peripheral Neuropathy, when in induction phase of their therapeutic protocol

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Pain scores | on average of 16 weeks
  Pain scores in the two treatment groups assessed at baseline and at the end of the treatment by age-appropriate pain scales. FLACC (the Faces, Legs, Arms, Cry and Consolability - pts aged 3-24 months) scale composed by 5 categories. Each category is scored on the 0-2 scale, which results in a total score of 0-10, where 0=Relaxed and comfortable, 4-6=Moderate pain, 1-3=Mild discomfort, 7-10=Severe discomfort or pain or both.
  FPS-R scale (Faces Pain Scale - Revised - pts aged 3-7 years): score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
  NRS-11(Numerical Rating Scale - pts aged 8-17 years): numerical rating scale where 0=no pain and 10=worst possible pain

SECONDARY OUTCOMES:
Percentage of responders to treatments | on average of 16 weeks
  Percentage of responders to treatments, defined as subjects with a pain intensity reduction of 30% from baseline. Pain intensity is evaluated using age-appropriate pain scale (FLACC, FPS-R, NRS-11).
  the FLACC (the Faces, Legs, Arms, Cry and Consolability- pts aged 3-24-months) scale is composed by 5 categories. Each category is scored on the 0-2 scale, which results in a total score of 0-10, where 0=Relaxed and comfortable, 4-6=Moderate pain, 1-3=Mild discomfort, 7-10=Severe discomfort or pain or both.
  FPS-R (Faces Pain Scale - Revised - pts aged 3-7 years) Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
  NRS-11 (Numerical Rating Scale - pts aged 8-17 years): numerical rating scale where 0=no pain and 10=worst possible pain.
Daily pain intensity | an average of 3 weeks
  Daily pain intensity, assessed by age-appropriate scale (FLACC, FPS-R or NRS-11) during dose optimization.
  the FLACC (the Faces, Legs, Arms, Cry and Consolability- pts aged 3-24-months) scale is composed by 5 categories. Each category is scored on the 0-2 scale, which results in a total score of 0-10, where 0=Relaxed and comfortable, 4-6=Moderate pain, 1-3=Mild discomfort, 7-10=Severe discomfort or pain or both.
  FPS-R (Faces Pain Scale - Revised - pts aged 3-7 years) Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
  NRS-11 (Numerical Rating Scale - pts aged 8-17 years): numerical rating scale where 0=no pain and 10=worst possible pain.
Observational assessment of pain | on average of 16 weeks
  Observational assessment of pain using the NRS-11 completed by parents and Investigator (or caregiver) at each visit.
  NRS-11 (Numerical Rating Scale): numerical rating scale where 0=no pain and 10=worst possible pain.
Self-assessment of pain for children ≥8 years of age | on average of 16 weeks
  Self-assessment of pain for children ≥8 years of age using the FPS-R pain scale at each visit.
  FPS-R (Faces Pain Scale - Revised) Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
Extent of pain | on average of 16 weeks
  Extent of pain evaluated as the number of painful areas using the pain charts at screening visit (V1), randomisation (v2) and EOS visit (V10).
  The pain charts are body maps (front and back) in which each body section is identified with a number.
Number of episodes of breakthrough pain | on average of 15 weeks
  Number of episodes of breakthrough pain (>7/10 pain score and use of rescue medications) during treatment period
Number of rescue interventions required during treatment period | on average of 15 weeks
  Number of rescue interventions required during treatment period.
Number of pain-free days | on average of 15 weeks
  Number of pain-free days (<4/10 average pain score without the use of rescue medications) during treatment period
Participant dropouts | up to 21 weeks
  Participant dropouts due to lack of adequate pain response.
The total cumulative weight normalized dose of each rescue drug. | on average of 16 weeks
  The total cumulative weight normalized dose of each rescue drug.
Total Summary Score from PedsQL™ scale | on average of 15 weeks
  Total score obtained using the PedsQL 4.0 Generic Core Scales (by parent, patient aged 3-17years) and PedsQL Infants Scales (by parent of pts aged 3-24months) at randomisation (V2) and at EOS (V10). The total score is a measure of Health Related Quality of life (HRQoL). Higher scores indicate better HRQOL.
  PedsQL 4.0 Generic Core Scales is composed by 4 multidimensional scales (Physical Funct, Emotional Funct, Social Funct, School Funct) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). Scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
  PedsQL Infant Scales is composed by 5 multidim. scales (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, Cognitive Functioning) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). The scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always)
Physical Health Summary Score from PedsQL™ scale | on average of 15 weeks
  Physical Health Score obtained using the PedsQL™ 4.0 Generic Core Scales (by parent, patient aged 3-17 years) and PedsQL™ Infant Scales (by parent, aged 3-24 months) at randomisation (V2) and at EOS (V10).
  PedsQL™ 4.0 Generic Core Scales is composed by 4 multidimensional scales (Physical Funct, Emotional Funct, Social Funct, School Funct) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). Scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
  PedsQL™ Infant Scales is composed by 5 multidimensional scales (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, Cognitive Functioning) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). The scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
Psychosocial Health Summary Score from PedsQL™ scale | on average of 15 weeks
  Psychosocial Health Score obtained using the PedsQL™ 4.0 Generic Core Scales (by parent, patient aged 3-17 years) and PedsQL™ Infant Scales (by parent, aged 3-24 months) at randomisation (V2) and at EOS (V10).
  PedsQL™ 4.0 Generic Core Scales is composed by 4 multidimensional scales (Physical Funct, Emotional Funct, Social Funct, School Funct) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). Scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
  PedsQL™ Infant Scales is composed by 5 multidimensional scales (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, Cognitive Functioning) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). The scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
Acceptability of treatment | at week 16
  Acceptability of treatment (Five Point Facial Hedonic Scale) at EOS visit (V10).
  Each face in the scale is related to a score (1=unpleasant; 2=not sure; 3=pleasant).
Global satisfaction with treatment | at week 16
  Global satisfaction with treatment (NRS-11, by parent, patient) at EOS visit (V10).
  The satisfaction is measeured by the numerical rating scale NRS-11 where 0=not satisfied and 10=fully satisfied
Clinical Global Impression of Severity of the subject's condition | an average of 15 weeks
  Clinical Global Impression of Severity (CGI-S) for Neuropathic or Mixed Pain Overall Severity Prior to Study Treatment (at randomization - V2) assessed by Investigator.
  Investigators will rate their impression of the severity of the subject's condition.
  Scoring: Normal: no signs of pain, Borderline painful, Mildly painful, Moderately painful, Markedly painful, Severely painful, Among the most extremely painful patients.
Clinical Global Impression of Improvement for pain | an average of 15 weeks
  Clinical Global Impression of Improvement (CGI-I) for Neuropathic or Mixed Pain Overall at V6 and EOS visit (V10) assessed by Investigator.
  Investigators will rate their impression of any change of the subject's overall condition of neuropathic or mixed pain since randomization in the study. Scoring are: Very much improved since the initiation of treatment; Much improved; Minimally improved; No change from baseline (the initiation of treatment); Minimally worse; Much worse; Very much worse since the initiation of treatment.
Patient/parent Global Impression of Change | an average of 12 weeks
  Patient/parent Global Impression of Change (PGIC; by parent, patient) at V6 and EOS visit (V10).
  Patient/parent will rate their impression of any change of the subject's overall condition of neuropathic or mixed pain since randomization in the study. Scoring are: Very much improved since the initiation of treatment; Much improved; Minimally improved; No change from baseline (the initiation of treatment); Minimally worse; Much worse; Very much worse since the initiation of treatment.
CL/F | at week 3 or at week 4 or at week 16
  Primary pharmacokinetic parameters for gabapentin: assessment of apparent clearance (CL/F) and of its variability and precision. In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Vd/F | at week 3 or at week 4 or at week 16
  Primary pharmacokinetic parameter for gabapentin: assessment of apparent volume of distribution (Vd/F) and of its variability and precision. In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
ka | at week 3 or at week 4 or at week 16
  Primary pharmacokinetic parameter for gabapentin: assessment of absorption rate constant (Ka) and of its precision and variability. In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
AUC | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin: assessment of Area under the Concentration curve (AUC). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Cmax | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin: assessment of peak plasma concentration (Cmax). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Tmax | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin: assessment of time at which the Cmax is observed (Tmax). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Css | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin: assessment of steady state Concentrations (Css). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Cmin | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin: assessment of minimum concentration (Cmin). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Systemic exposure to investigational product | an average of 12 weeks
  Systemic exposure to investigational product during maintenance period, as assessed by predicted steady-state concentrations.
Incidence of Adverse Events | up to 21 weeks
  Incidence of Adverse Events at all visits
Percentage of subjects discontinuing the Trial | up to 21 weeks
  Percentage of subjects discontinuing the Trial due to treatment-emergent adverse events
Aggressive behaviour in children aged >6 years | an average of 15 weeks
  Aggressive behaviour in children aged >6 years using the Retrospective Modified Overt Aggression Scale (R-MOAS) at V2, V6 and EOS visit (V10).
  The scale includes 4 domains (Verbal Incidents, Incidents Toward Other People, Incidents Involving Property, Incidents Directed Toward Self) each one describing different behaviours.
  Parents rate the frequency of 16 aggressive behaviors (referred to the past week) in the 4 areas. Numeric weighting amplifies the seriousness of more harmful behaviors in the total score. Higher score indicating more aggressive behavior.
Suicidal ideation/behaviour in subjects aged 6 years and older | an average of 16 weeks
  Suicidal ideation/behaviour in subjects aged 6 years and older using the Columbia - Suicide Severity Rating Scale (C-SSRS) scores before IMP (screening V1), V6, EOS visit (V10) and taper visit (V11).
  The C-SSRS is divided into 2 sections: Suicidal Ideation and Suicidal Behaviour containing each one 5 "yes" or "no" questions.
  Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. A score of 0 is assigned if no ideation is present.
  Composite endpoints are defined below:
  Suicidal ideation: A "yes" answer at any time during treatment to any one of the five suicidal ideation questions (Categories 1-5).
  Suicidal behavior: A "yes" answer at any time during treatment to any one of the five suicidal behavior questions (Categories 6-10).
  Suicidal ideation or behavior: A "yes" answer at any time during treatment to any one of the ten suicidal ideation and behavior questions (Categories 1-10)
Assessment of blinding | at week 16
  Assessment of blinding: guess of the subject's treatment group (by Investigator, parents and subject if at adequate maturity level) at V10.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia De Wildt, MD-PhD, Principal Investigator — Erasmus Medical Center

REFERENCES:
- [Background] Finnerup NB, Sindrup SH, Jensen TS. Recent advances in pharmacological treatment of neuropathic pain. F1000 Med Rep. 2010 Jul 14;2:52. doi: 10.3410/M2-52. PMID 21170362
- [Background] Mellegers MA, Furlan AD, Mailis A. Gabapentin for neuropathic pain: systematic review of controlled and uncontrolled literature. Clin J Pain. 2001 Dec;17(4):284-95. doi: 10.1097/00002508-200112000-00002. PMID 11783808
- [Derived] de Leeuw TG, Mangiarini L, Lundin R, Kaguelidou F, van der Zanden T, Pasqua OD, Tibboel D, Ceci A, de Wildt SN; GAPP consortium. Gabapentin as add-on to morphine for severe neuropathic or mixed pain in children from age 3 months to 18 years - evaluation of the safety, pharmacokinetics, and efficacy of a new gabapentin liquid formulation: study protocol for a randomized controlled trial. Trials. 2019 Jan 15;20(1):49. doi: 10.1186/s13063-018-3169-3. PMID 30646965
- See also: The Task force in Europe for Drug Development for the Young (TEDDY) is a network of excellence funded in 2005 as a consortium responding to a call published by the European Commission. — http://www.teddynetwork.net/